CLINICAL TRIAL: NCT01528969
Title: The Effect of the Frequent Xylitol Chewing Gum Use on the Oral Microbiota in Children With High MS Counts
Brief Title: Effect of Xylitol on Oral Microbiota in Children
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kuwait University (Other)
Collaborators: University of Turku (Other); University of Michigan (Other)
Responsible Party: Principal Investigator, Eino Honkala, Professor, Kuwait University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DD02/10; KU-DD02/10 (Other Grant/Funding Number: Kuwait University)
Record Dates: First submitted 2012-01-24; First posted 2012-02-08 (Estimated); Results first posted 2015-08-10 (Estimated); Last update posted 2015-08-10 (Estimated); Status verified 2015-07

CONDITIONS: Bacterial Infections
Keywords: oral microbiota; mutans streptococci; xylitol
MeSH Terms: conditions — Bacterial Infections | interventions — Xylitol; Sorbitol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Xylitol (Experimental): A half of the subjects will be randomly allocated into xylitol group.
  Interventions: Dietary Supplement: xylitol
- Sorbitol (Active Comparator): About 40 randomly allocated subjects will chew sorbitol chewing gum (1,5, g/pellet) three times a day
  Interventions: Dietary Supplement: sorbitol

INTERVENTIONS:
Dietary Supplement: xylitol — Subjects will chew 2 pieces of xylitol chewing gum (1,5 g/pellet) three times a day in the experimental group for a five-week period.
  Other Names: Xylitol chewing gum; Sorbitol chewing gum
  Arms: Xylitol
Dietary Supplement: sorbitol — Subjects will chew 2 pieces of sorbitol chewing gum (1,5 g/pellet) three times a day in the control group for a five-week period.
  Other Names: Sorbitol chewing gum
  Arms: Sorbitol

SUMMARY:
1. The present controlled, randomized, doubleblind study aims to answer the following questions:

   * How will the "normal flora" be affected by the xylitol consumption?
   * Will daily consumption of xylitol change the plaque-saliva distribution of the mutans streptococci?
   * The association of the test results will also be compared with the caries status at the baseline.
2. About eighty subjects with MS counts of log CFU 5 or more will be identified and invited to the study. They will be randomly divided into a Xylitol and Sorbitol group.
3. Xylitol/Sorbitol gum (6g polyol/day) will be used for 5 weeks. Saliva samples will be collected before and after gum use.
4. Studying and quantifying of 16 bacterial species belonging to the normal flora by DNA-DNA hybridizations and Real-time PCR will show how xylitol influenced the oral flora in general.

DETAILED DESCRIPTION:
Xylitol, a 5-carbon polyol, has in clinical studies prevented caries occurrence in children and decreased counts of mutans streptococci (MS) and the amount of plaque when used on daily basis. How xylitol influences mutans streptococci is far from clear. Also the effects of xylitol on the normal flora are poorly understood.

The present controlled, randomized, doubleblind study aims to answer the following questions:

1. How will the "normal flora" be affected by the xylitol consumption?
2. Will daily consumption of xylitol change the plaque-saliva distribution of the mutans streptococci?
3. The association of the test results will also be compared with the caries status at the baseline.

After collecting informed consent forms from the parents, about 177 children will be screened for the presence of salivary mutans streptococci (SM) with chairside test, Dentocult SM® Strip mutans (Orion Diagnostica, Finland).

Sorbitol is regarded as an inert polyol. Xylitol/Sorbitol gum (6g polyol/day) will be used for 5 weeks. Saliva samples will be collected before and after gum use. Studying and quantifying of 16 bacterial species belonging to the normal flora by DNA-DNA hybridizations and Real-time PCR will show how xylitol influenced the oral flora in general. Comparison of MS counts in unstimulated vs. stimulated saliva will show how xylitol affected the adhesivity of the MS.

ELIGIBILITY:
Inclusion Criteria:

* high SM count

Exclusion Criteria:

* low SM count,
* ongoing medication

Ages: 11 Years to 14 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 122 (Actual)
Dates: Start 2012-03; Primary Completion 2012-04 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eino Honkala, PhD, Principal Investigator — Faculty of Dentistry, Kuwait University
Locations (1):
- Faculty of Dentistry, Kuwait University, Kuwait City, Kuwait

REFERENCES:
- [Background] Honkala E, Honkala S, Shyama M, Al-Mutawa SA. Field trial on caries prevention with xylitol candies among disabled school students. Caries Res. 2006;40(6):508-13. doi: 10.1159/000095650. PMID 17063022
- [Background] Honkala E, Rimpela A, Karvonen S, Rimpela M. Chewing of xylitol gum--a well adopted practice among finnish adolescents. Caries Res. 1996;30(1):34-9. doi: 10.1159/000262134. PMID 8850581

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Altogether 122 10-12-year-old boys, whose parents gave a positive consent, participated in the baseline examinations. The study was conducted at one school in Jabriya, Kuwait.
Pre-assignment Details: Str mutans was measured from plaque and saliva. Those children who had high mutans counts (n=75) were included into the intervention.
Groups:
- Xylitol: A half of the subjects (n = 37) were randomly allocated into xylitol group.
  Subjects chewed 2 pieces of xylitol chewing gum (1,5 g/pellet) three times a day for five weeks.
- Sorbitol: A half of the subjects (n = 38) were randomly allocated into sorbitol group.
  Subjects will chewed 2 pieces of sorbitol chewing gum (1,5, g/pellet) three times a day for five weeks.
Period: Overall Study
Arm/Group | Xylitol | Sorbitol
Started | 37 | 38
Completed | 35 | 38
Not Completed | 2 | 0
Not completed — absent from the school at baseline | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Xylitol: A half of the subjects (n = 37) were randomly allocated into xylitol group.
  Subjects chewed 2 pieces of xylitol chewing gum (1,5 g/pellet) three times a day for five weeks. Each chewing gum pellet contained 65% xylitol w/w.
- Sorbitol: A half of the subjects (n = 38) were randomly allocated into sorbitol group.
  Subjects will chewed 2 pieces of sorbitol chewing gum (1,5, g/pellet) three times a day for five weeks. Each chewing gum pellet contained sorbitol 63% and sorbitol 2%.
- Total: Total of all reporting groups
Arm/Group | Xylitol | Sorbitol | Total
Number analyzed (Participants) | 37 | 38 | 75
Age, Continuous [Mean (Full Range); unit: years] | 11.5 [10 to 12] | 11.5 [10 to 12] | 11.5 [10 to 12]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 37 | 38 | 75
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 37 | 38 | 75
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 37 | 38 | 75
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Kuwait | 37 | 38 | 75
Nationality of subjects [Number; unit: participants]
  Kuwaiti | 36 | 37 | 73
  non-Kuwaiti Arab | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: MS Counts of Stimulated Saliva
Description: The MS counts were measured at the beginning and in the end of the 5 weeks intervention
Time Frame: 5 weeks
Measure: Mean (Standard Deviation); unit: MS counts log CFU/ml
Arm/Group | Xylitol | Sorbitol
Number analyzed (Participants) | 35 | 38
MS counts log CFU/ml
  Baseline | 4.86 (1.34) | 4.40 (1.71)
  5-week follow-up | 4.29 (1.73) | 3.78 (1.83)

2. Secondary Outcome: The Changes in the Counts of the 14 Other Bacterial Species
Description: The bacterial species were measured from stimulated saliva at the beginning and after the intervention
Time Frame: 5 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: during the 1st week after the intervention was concluded.
Description: Subjects were interviewed about the possible side-effects (e.g. diarrhea) after the five-weeks intervention in the connection of the follow-up examinations.
Groups:
- Xylitol: A half of the subjects (n = 37) were randomly allocated into xylitol group.
  Subjects chewed 2 pieces of xylitol chewing gum (1,5 g/pellet) three times a day for five weeks. Each chewing gum pellet contained 65% xylitol w/w.
  None of the subjects had any adverse effects of the consumption of the chewing gum.
- Sorbitol: A half of the subjects (n = 38) were randomly allocated into sorbitol group.
  Subjects will chewed 2 pieces of sorbitol chewing gum (1,5, g/pellet) three times a day for five weeks. Each chewing gum pellet contained sorbitol 63% and sorbitol 2%.
  None of the subjects had any adverse effects of the consumption of the chewing gum.
Arm/Group | Xylitol | Sorbitol
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/38
Other Adverse Events (participants affected / at risk) | 0/35 | 0/38
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Xylitol (N=35) | Sorbitol (N=38)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) — Interview after the intervention

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes